CLINICAL TRIAL: NCT06371495
Title: Statins in Acute Ischemic Stroke(Role of Statins in Reperfusion in Acute Stroke )
Brief Title: Statins Role in Acute Ischemic Stroke
Acronym: observation
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Mohamed Sedeq, Dr, Assiut University
Other Study IDs: statins in ischemic stroke
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group ABC: GroupA: recieve rosuvastatin 40mg
  Interventions: Drug: rosuvastatin
- Group B: Group B :recive rosuvastatin20
  Interventions: Drug: rosuvastatin

INTERVENTIONS:
Drug: rosuvastatin — Stude include three groupsof people GroupA: recieve rosuvastatin 40mg Group B :recive rosuvastatin 20mg Group C: recive placebo 2- Follow up will be done using NIHSS at the onset and modified Rankin scale at the onset and after 1 month and 3 months of the onset.
  3- Carotid duplex will be done at the onset and after 1 month and 3 months of the onset.
  Other Names: ststins

SUMMARY:
Strokes is amajor cause of death and disabilities in different countried

DETAILED DESCRIPTION:
Stroke is a major cause of mortality and disability in modern societies. Statins are effective medications in decreasing cardiovascular events through lipid lowering and pleiotropic effects. Ischemic stroke is burdened with a high morbidity and mortality in our society. However, there are few effective and largely available therapies for this devastating disease. In additon to advancing acute reperfusion therapies, there is a need to develop treatments aimed to promote repair and regeneration of brain tissue damaged by ischemia (neurorecovery)(1,2,3). Therapeutic angiogenesis and vasculogenesis represent novel approaches of regenerative medicine that may help in the cure of patients with acute ischemic stroke. Translation of our knowledge about these processes from the bench to bedside is still underway. Although angiogenesis (the sprouting of new blood vessels from pre-existing vascular structures) is likely to contribute to neurorepair, the finality of the angiogenic response in acute ischemic stroke has not been fully elucidated. The first therapeutic approach to angiogenesis after ischemic stroke would be the modulation of the endogenous angiogenic response. In this setting, early instauration of physical activity, statins, and peroxisome proliferator-activated receptor-γ agonists may enhance angiogenesis and neuroregeneration Statins have been shown to improve the functional outcome of patients after an ischemic stroke. We hypothesized that daily statin intake improves functional outcome after an acute ischemic stroke (4,5,6,7,8) Duplex sonography is the best noninvasive modality for investigation of possible carotid artery stenosis to evaluate the intema media thickness of carotid artery in patients of acute ischemic stroke before and after receiving high dose of statins to evaluate its effectiveness in management and appropriate dose of statins (9.10.11.12,13,14)

ELIGIBILITY:
Inclusion Criteria:

* .patients.have acute ischemic stroke within 24 hours of onset. 2.patient not received intravenous thrombolysis or mechanical thrombectomy3.patients with no contraindications or hypersensitivity to statins

Exclusion Criteria:

* 1. Patient received IV thrombolysis or underwent mechanical thrombectomy 2. patient have acute ischemic stroke with onset of more than 24 hours 3.patients have hypersestivty or contraindication to statin 4:patients refuse to participate in the study

Ages: 20 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: people have acute ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2024-08-13 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Carotid duplex will be done at the onset and after 1 month and 3 months of the onset. | first day and after 3 mounths
  measure the carotid thickness through Carotid duplex

REFERENCES:
- [Result] Gandhi BS, Kanungo MS. Effect of cortisone on monoamine oxidase of the liver of young & old rats. Indian J Biochem Biophys. 1974 Jun;11(2):102-4. No abstract available. PMID 4448456